CLINICAL TRIAL: NCT00899418
Title: Differential Response of Breast Cancer Patients on E2100 Treated With Bevacizumab as a Function of Genetic Polymorphisms of VEGF and KDR
Brief Title: Studying Tumor Tissue Samples to Learn More About DNA Changes and Response in Patients With Breast Cancer Treated With Bevacizumab on Clinical Trial ECOG-2100
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000472065; U10CA021115 (NIH); ECOG-E2100T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2008-10

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This laboratory study is examining tumor tissue samples from patients with breast cancer treated with bevacizumab on clinical trial ECOG-2100 to learn more about DNA changes and response in these patients.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the effect of known variant polymorphisms (with functionally important associations) of the vascular endothelial growth factor (VEGF) gene on outcome (time to progression) in patients with breast cancer treated with bevacizumab on clinical trial ECOG-2100.

Secondary

* Assess the effect of known variant polymorphisms (with functionally important associations) of the VEGF receptor-2 (KDR) gene on outcome (time to progression) in these patients.
* Assess the effect of known variant polymorphisms of these genes on efficacy (objective response rate and survival) in these patients.
* Assess the effect of known variant polymorphisms of these genes on toxicity outcome in these patients.
* Assess the effect of VEGF polymorphisms on VEGF expression by immunohistochemical staining (a known prognostic marker).
* Assess the effect of KDR polymorphisms on KDR expression by immunohistochemical staining.

OUTLINE: This is a multicenter study.

Tissue and genomic DNA samples from paraffin-embedded primary tumor are examined using standard polymerase chain reaction (PCR) restriction fragment-length polymorphisms, immunohistochemistry, allele-specific PCR, and/or Taqman-based assays. Vascular endothelial growth factor (VEGF) and VEGF receptor-2 (KDR) expression and polymorphisms are assessed.

PROJECTED ACCRUAL: A total of 500 specimens will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast
* Enrolled on clinical trial ECOG-2100 and received treatment with bevacizumab
* Paraffin-embedded tumor samples available
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Time to progression in patients with a known polymorphism vs those with wild-type vascular endothelial growth factor (VEGF) gene

SECONDARY OUTCOMES:
Time to progression in patients with a known polymorphism vs those with wild-type VEGF receptor-2 (KDR) gene
Difference in response rate, survival, and toxicity in patients with a known polymorphism vs wild-type VEGF and KDR

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P. Schneider, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center